CLINICAL TRIAL: NCT06333834
Title: Assessment of the Efficacy of Anti-scorpion Venom Therapy in a Dose-response Manner, Following the Principles of Rational Drug Use in Patients With Scorpionism: a Non-inferiority, Randomized, Double-blind, Controlled Clinical Trial
Brief Title: Assessment of the Efficacy of Scorpion Antivenom Therapy in a Dose-response Manner, in Patients With Scorpionism
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Selene Guadalupe Huerta Olvera (Other)
Responsible Party: Sponsor-Investigator, Selene Guadalupe Huerta Olvera, Professor and researcher, University of Guadalajara
Organization: University of Guadalajara (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Dosis Seriada de Alacramyn
Record Dates: First submitted 2024-03-05; First posted 2024-03-27 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Centruroides Envenomation
Keywords: Centruroides; Antivenom; Scorpion antivenom; Scorpion envenomation
MeSH Terms: conditions — Scorpion Stings

STUDY DESIGN:
Intervention Model Description: Experimental Group: Patients with scorpion envenomation of any grade will receive scorpion antivenom therapy in a reduced regimen. The dosing regimen based on response will be one initial intravenous vial in patients with grade III scorpion envenomation, and two initial intravenous vials as the starting dose in patients with grade IV scorpion envenomation, according to the FDA classification of scorpion envenomation. In both scenarios, an additional vial can be administered every 30 minutes if symptoms persist, with no limit on vials. Control Group: Patients with scorpion envenomation of any grade will receive scorpion antivenom therapy according to the traditional regimen proposed in the Mexican Clinical Practice Guideline, where, according to the severity classification of scorpion envenomation, between one and six vials of anti-scorpion venom will be administered, and equal doses can be repeated every 30 minutes if necessary.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A pharmacist will be responsible for randomizing the patients and preparing the study medication in a blinded manner, so that the treatment is administered by the physician without the care provider or the participant being able to identify it. The pharmacist will keep the randomization results in a sealed envelope that will be opened at the end of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Traditional scorpion antivenom regimen (Active Comparator): Active/placebo comparator
  Interventions: Drug: Traditional scorpion antivenom regimen
- Serial dose of scorpion antivenom regimen (Experimental)
  Interventions: Drug: Serial dose of scorpion antivenom regimen

INTERVENTIONS:
Drug: Traditional scorpion antivenom regimen — All patients will be classified according to two severity scales. The pharmacist, who is the only team member aware of which group each patient was assigned to, will consider the classification corresponding to the classification proposed by the Mexican Clinical Practice Guideline to decide the dose of scorpion antivenom. Scorpion antivenom will be administered to all patients. Patients in this group will receive between one and three vials every 30 minutes, depending on the severity of the condition (one vial for patients classified as grade I, two vials for patients classified as grade II, and three vials for patients classified as grade III)
  Arms: Traditional scorpion antivenom regimen
Drug: Serial dose of scorpion antivenom regimen — All patients will be classified according to two severity scales. The pharmacist, who is the only team member aware of which group each patient was assigned to, will consider the classification corresponding to the American classification to decide the dose of scorpion antivenom. Scorpion antivenom will be administered only in the presence of signs and/or systemic symptoms of intoxication, excluding signs and symptoms at the sting site. Patients in this group will receive between one and two vials every 30 minutes, depending on the severity of the condition (one vial for patients classified as grade III and two vials for patients classified as grade IV)
  Arms: Serial dose of scorpion antivenom regimen

SUMMARY:
The clinical study aims to compare the effectiveness of applying two different regimens of scorpion antivenom therapy. In the first regimen (control), the medication is administered to all patients, and depending on the severity of the condition, the dosage varies. In the experimental regimen, an identical dose of scorpion antivenom is administered to patients exhibiting signs and symptoms of scorpion sting intoxication, in addition to pain and other symptoms at the sting site. The primary response variable is the time taken for signs and symptoms to resolve, but differences in complications, adverse effects, venom and antivenom concentration in the blood, and the need for other therapeutic measures are also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 or older presenting with a diagnosis of scorpionism to the emergency department.
* Treated solely with paracetamol, scorpion antivenom, saline solution, and local ice application.
* Any gender.
* Less than two hours elapsed since scorpion sting.
* Willing to participate in the study through written informed consent.

Exclusion Criteria:

* Allergies or contraindications to any of the study medications.
* Uncertainty regarding scorpion sting.
* Previous treatment by another physician.
* Intramuscular administration of scorpion antivenom due to urgent clinical conditions.
* Decision not to provide informed consent.
* Any limitations hindering the proper understanding of study participation.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2024-06-15 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Time to resolution of signs and symptoms | two and a half to five hours
  Time to resolution of signs and symptoms from admission and from the estimated time of the sting
Serum venom concentration | two and a half to five hours
  Serum venom concentration upon patient arrival, after administration of antivenom, and upon reporting the absence of signs of intoxication

SECONDARY OUTCOMES:
Mortality | two and a half to five hours
  Mortality rate of each group
Length of intrahospital stay | two and a half to five hours
  Time from patient admission to discharge due to patient improvement
Serum antivenom concentration | two and a half to five hours
  Scorpion antivenom concentration at five minutes after administration, prior to secondary doses, and prior to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Selene G Huerta-Olvera, PhD, Study Director — Medical & Life Sciences Department. La Ciénega University Center; Héctor A González-Ruiz, PhD student, Principal Investigator — Centro Universitario de Ciencias de la Salud
Locations (1):
- Servicios Médicos Municipales de San Pedro Tlaquepaque., Tlaquepaque, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ziggelaar A. [The origin of the theory of harmonious vibrations. The father, Ignace Gaston Pardies (1636-1673). Studies on Ignace gaston Pardies I]. Dent Mag Oral Top. 1966 Apr;83(2):145-51. No abstract available. French. PMID 5330957